CLINICAL TRIAL: NCT03609788
Title: Validation of the Turkish Version of the Pain Sensitivity Questionnaire in Patients With Chronic Pain
Brief Title: Validation of the Turkish Version of the Pain Sensitivity Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ferda Yilmaz Inal, Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 71306642-050.01.04-10/12
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Pain
Keywords: pain sensitivity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Pain Sensitivity Questionnaire(PSQ) is a self-rating measure for the assessment of pain sensitivity and has been developed by Dr. R. Ruscheweyh in Germany. It consists of 17 items rated from 0, not at all painful to 10, most severe pain imaginable. The validation of the Turkish version of PSQ is needed, in order to measure pain sensitivity among Turkish people.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* adult chronic low back pain patients having pain for greater than 3 months

Exclusion Criteria:

* Failed back surgery syndrome,
* Morbid obesity (body mass index, >40),
* Being a non-Turkish speaker,
* Substance abuse disorder,
* Major psychiatric disorder (eg, severe depression, bipolar disorder, Axis II personality disorder, and schizophrenia).

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo a low back interventional procedure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of pain intensity in Turkish people using The Turkish version of the PSQ | 1 day
  Measurement of pain intensity in Turkish people using The Turkish version of the PSQ, consisting of 17 items, describing different daily life situations with a scoring from 0(not painful) to 10 (worst pain imaginable) on a numeric rating scale. A PSQ total score is between 0-10, the higher score, the more patient's pain sensitivity.
Pain Catastrophizing Scale | 1 day
  This scale is used in order to assess the state of mind of patients in pain through a comprehensive evaluation instrument that encompasses the different perspectives on catastrophizing. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52.24 The higher the score, the more catastrophizing thoughts are present.
Beck Anxiety Inventory | 1 day
  This scale, consisting of 21 items, is a self-report measure of anxiety. Score of 0-21 shows low anxiety. Score of 22-35 shows moderate anxiety. Score of 36 and above shows potentially concerning levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)